CLINICAL TRIAL: NCT06009679
Title: MISOPROSTOL FOR THE TREATMENT OF SUSPECTED POSTPARTUM RETAINED PRODUCTS OF CONCEPTION - A RANDOMIZED TRIAL
Brief Title: MISOPROSTOL FOR THE TREATMENT OF SUSPECTED POSTPARTUM RETAINED PRODUCTS OF CONCEPTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Principal Investigator, Oshri Barell, DR OSHRI BAREL, Assuta Ashdod Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000621AAA
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Retained Products of Conception
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: Two arms: the intervention groups will include patients with suspected postpartum RPOC that will receive treatment with Misoprostol, and the control group will undergo conservative follow-up with ultrasound. The primary endpoint will be the number of patients with histopathology-proven retained products of conception at 8-16 weeks postpartum in each group. secondary endpoints will be the number of hysteroscopies in each group, side effects of treatment, late postpartum hemorrhage, blood transfusion, endomyometritis / PID and re-admissions to the hospital in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will include patients with suspected postpartum RPOC that will receive treatment with Misoprostol, 600 microgram SL/PO/PV
  Interventions: Drug: Misoprostol 200mcg Tab
- Control group (No Intervention): The control group will include women with suspected postpartum RPOC per ultrasound examination that will undergo conservative follow-up with ultrasound for a period of 6-12 weeks postpartum

INTERVENTIONS:
Drug: Misoprostol 200mcg Tab — Patients in the intervention group with suspected postpartum RPOC will receive 600 micrograms of misoprostol up to 3 times following delivery and followed up by ultrasound and clinical examinations for 6-12 weeks post-partum
  Arms: Intervention group

SUMMARY:
The goal of this current study is to evaluate the efficacy of treatment of postpartum patients with suspected retained products of conception (RPOC) with Misoprostol in reducing the frequency of postpartum RPOC compared to a control group of patients that will be managed expectantly, in a prospective randomized trial.

DETAILED DESCRIPTION:
Misoprostol (Cytotec) is used widely in Obstetrics and Gynecology, whether for labor induction (1), prevention (2), and treatment (3) of early postpartum hemorrhage (ePPH), induced and missed abortions (4) and for cases suspected for having retained products of conception postabortion and postpartum (RPOC, residua).

While it has been shown in previous studies that misoprostol is efficacious for most of the above-mentioned indications, it is less well-established that the treatment for suspected postpartum RPOC alters the natural course of events and reduces the number of patients requiring surgical intervention and actually having RPOC.

RPOC is estimated to complicate about 1% of term pregnancies and is more prevalent than after miscarriages and termination of pregnancy (5).

The diagnosis and treatment of RPOC might be challenging, as there are no clearly determined diagnostic criteria, evidence-based guidelines or treatment protocols (6).

Different protocols for the follow-up and treatment of cases suspected of RPOC are in use worldwide, including expectant management, administrating uterotonics, performing suction curettage (6), and performing hysteroscopy (7, 8). Evidence in the literature supports the treatment of RPOC with operative hysteroscopy since curettage seems to increase the risk for intrauterine adhesions and Asherman syndrome (9, 10) with the possibility for menstrual abnormalities, infertility or subfertility, recurrent pregnancy losses, preterm labor, and preterm premature rupture of membranes (11).

Chambers et al published in 2009 a 6-year trial (12), which shows that treatment with 200 mcg SL / PO misoprostol 3 times daily for 2 days may effectively treat RPOC and reduce repeat curettage rate by 79.6%. There was also the complete resolution of symptoms in 93%, and 77% of women reported a high level of satisfaction. The trial was retrospective and RPOC was not confirmed by hysteroscopy or histology.

The main tool for diagnosis and follow-up in cases of RPOC is postpartum ultrasound, showing low, medium, and high probability for residua, with the clinical symptoms of abnormal bleeding pattern, abdominal tenderness, and persistently dilated cervix.

We've decided to set the categories according to the study by Smorgick (13), although we chose to name them and treat them differently. The categories are:

1. Low probability for residua - ultrasound shows thin regular endometrial line 10 mm and below, with no intrauterine mass or Doppler vascular flow.

   In effect a normal ultrasound scan.
2. Medium probability for residua - ultrasound shows a cavity over 10 mm, intrauterine hypo / hyperechogenic mass, or irregular endometrial line without Doppler flow. With this group, PROC cannot be excluded.
3. High probability for residua - with the addition of Doppler vascular flow to the cavity.

The natural course of the ultrasonic appearance of the uterine cavity postpartum (14) was shown to take roughly 56 days for the cavity to appear empty in 95% percent of cases not suspected of having RPOC.

This study aims to test prospectively expectant management compared to misoprostol administration for a certain duration of time of cases with risk factors for RPOC, including cases undergoing revision of the uterine cavity or manual lysis of placenta postpartum, early postpartum hemorrhage, cases with a history of treated postpartum residua, having placental pathology (succenturiate, bilobed placenta), a pregnancy that started as multifetal with only one fetus reached advanced pregnancy, and patients undergoing Bumm curettage post-delivery.

2. Aims Since the literature data on this subject is scarce and the treatment is challenging, the primary aim of this study is to assess prospectively and randomly expectant management vs. misoprostol administration (PV, PO, SL) on the treatment for suspected RPOC postpartum in women with risk factors for residua along an 8-week duration as characterized by ultrasound follow-up every 2-3 weeks and divided to a 3 tier system of the low, medium and high probability of residua and the cases requiring hysteroscopy for suspected residua.

Secondary aims include side effects of treatment, late postpartum hemorrhage, blood transfusion, and endomyometritis / PID and complications.

3. Hypothesis In this study, we hypothesize that the treatment with misoprostol, compared to expectant management, will be able to reduce the number of cases at medium and high probability of residua as described by ultrasound and by that reduce the number of cases requiring hysteroscopy and treatment of residua.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 years - 45 years.
* Spontaneous vaginal delivery or vacuum extraction, including VBAC cases
* Revision of the uterine cavity or manual lysis of the placenta postpartum
* Early postpartum hemorrhage
* Cases with a history of treated postpartum residua (by curettage or hysteroscopy)
* Placental pathology (succenturiate placenta, bilobed placenta)
* Pregnancy that started as a multifetal gestation with only one fetus reached advanced pregnancy
* Bumm curettage post-delivery
* Patients are able to provide written consent

Exclusion Criteria:

* Patients with no risk factors of RPOC
* Cesarean section on index pregnancy
* Cases requiring urgent curettage for late postpartum hemorrhage
* Inability to consent due to cognitive or language barrier

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Cases of retained products of conception | 8-16 weeks postpartum
  The primary endpoint will be the number of patients with histopathology-proven retained products of conception at 8-16 weeks postpartum in each group.

SECONDARY OUTCOMES:
Need for hysteroscopy due to suspected RPOC | 8-16 weeks postpartum
  number of hysteroscopies in each group
side effects of treatment | 8-16 weeks postpartum
  any side effects of treatments with Misoprostol
Late postpartum hemorrhage | 6 weeks postpartum
  Late postpartum hemorrhage during the followup
Blood transfusions | 6-18 weeks postpartum
  The need of blood transfusion during the followup
endomyometritis / PID | 6-18 weeks postpartum
  any events of endomyometritis / PID postpartum
Re-admissions to the hospital | up to 18 weeks
  cases that required re-admission to the hospital after discharge from tyhe postpartum ward.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Ashdod University Hospital, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No